CLINICAL TRIAL: NCT01424592
Title: Inpatient Portable Sleep Apnea Testing of Hospitalized Medical Patients for the Evaluation of Obstructive Sleep Apnea Prospectively Compared to Outpatient Laboratory-based Polysomnography
Brief Title: In-Hospital Portable Sleep Monitoring for the Evaluation of Obstructive Sleep Apnea (OSA)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Swamy Nagubadi, Attending Physician: Pulmonary, Critical Care, and Sleep Medicine, Cook County Health
Other Study IDs: CCHHS IRB 11-027
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: Portable sleep apnea testing; Positive airway pressure therapy; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: Hospitalized inpatients referred by a general medicine service for evaluation of obstructive sleep apnea.
  Interventions: Device: Testing with a portable sleep apnea monitor .

INTERVENTIONS:
Device: Testing with a portable sleep apnea monitor . — Portable sleep apnea testing will performed on referred patients.
  Other Names: Alice PDx portable sleep testing system (Philips Respironics, Murraysville, PA)

SUMMARY:
Hypothesis: Portable sleep testing of hospitalized medical inpatients suspected of having OSA is accurate in determining the need for positive airway pressure (PAP) therapy when compared to outpatient laboratory-based polysomnography.

* Hospitalized medical inpatients referred for suspected OSA will be tested with a portable sleep apnea testing device during hospitalization.
* These patients will then undergo an outpatient laboratory-based attended polysomnography after hospital discharge.
* Results of the inpatient portable sleep apnea test will be compared to the outpatient laboratory-based polysomnography in terms of diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

- Hospitalized inpatients referred for evaluation of suspected obstructive sleep apnea

Exclusion Criteria:

* Patients admitted to surgical or obstetrics/gynecology services
* Patients with certain medical conditions (altered mental status not related to respiratory failure, septicemia, unstable psychiatric disorder, narcotic abuse and prior diagnosed sleep apnea)
* Patients with certain social histories (prisoners)
* Patients unable to use CPAP (facial deformity and traumatic facial injuries).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital under the general medicine service referred for evaluation of suspected obstructive sleep apnea.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2011-04; Primary Completion 2022-06 (Estimated); Study Completion 2024-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Swamy Nagubadi, MD, Principal Investigator — Attending Physician, Pulmonary, Critical Care and Sleep Medicine; Aiman Tulaimat, MD, Study Chair — Attending Physician, Pulmonary, Critical Care and Sleep Medicine; Rohit Mehta, MD, Study Director — Fellow Physician, Pulmonary, Critical Care and Sleep Medicine
Locations (1):
- John H Stroger Hospital of Cook County, Chicago, Illinois, United States

REFERENCES:
- [Result] Nagubadi S, Mehta R, Abdoh M, Nagori M, Littleton S, Gueret R, Tulaimat A. The Accuracy of Portable Monitoring in Diagnosing Significant Sleep Disordered Breathing in Hospitalized Patients. PLoS One. 2016 Dec 19;11(12):e0168073. doi: 10.1371/journal.pone.0168073. eCollection 2016. PMID 27992566